CLINICAL TRIAL: NCT02428686
Title: Treatment of Anemia With Epoetin Beta in Low Risk Myelodysplastic Syndrome With Analysis of the Impact on Quality of Life and Functional Capacity of Patients
Brief Title: Treatment of Anemia With Epoetin Beta in Low Risk Myelodysplastic Syndrome (MDS)
Acronym: EPO-QoL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Groupe Francophone des Myelodysplasies (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GFM EPO QoL
Record Dates: First submitted 2011-11-24; First posted 2015-04-29 (Estimated); Last update posted 2015-04-29 (Estimated); Status verified 2015-04

CONDITIONS: Myelodysplastic Syndromes
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — epoetin beta

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- epoetin beta (Experimental)
  Interventions: Drug: Epoetin beta (NeoRecormon)

INTERVENTIONS:
Drug: Epoetin beta (NeoRecormon) — Epoetin beta 60 000 IU/week
  Other Names: NeoRecormon

SUMMARY:
Chronic anemia is the symptom most frequently found at diagnosis in low risk myelodysplastic syndrome. It generates an increased rate of morbidity and mortality in this population of patients whose median age is high and the rate of co-mobidities important. The historical treatment is limited to transfusion support with a significant impact on quality of life and the incidence of secondary haemosiderosis, which contributes to the emergence of co-morbidities, especially cardiovascular. Treatment with rHuEPO allows for overall erythroid response in 40-60% of patients treated.

In this trial, the investigators intend to study the interest of a treatment with epoetin beta in patients with anemia <10 g / dL in the context of a myelodysplastic syndrome with IPSS score <1.

In addition to studying the erythroid response, the investigators will measure the impact on quality of life and functional performance.

Patients will receive epoetin beta (60 000UI/week). Response will be assessed after 12 and 24 weeks of treatment.

DETAILED DESCRIPTION:
Objective of the trial Assess the level of haematological response according to IWG 2000 and IWG 2006 criteria with a pattern of administration of high doses epoetin beta (NeoRecormon ®) for 12 and 24 weeks of treatment;

To evaluate the predictive value of the rate of reticulocytes at Day 8 on the erythroid response;

* Assess time to response
* Assess tolerance
* Assess the impact on quality of life using the FACT-An and EQ-5D measurement scales;
* Assess functional capacity:

Cardiovascular performance on effort by the 6-minute walk test Performing the " Short Physical Performance Battery " tests

Evaluation The evaluation of response according to the IWG 2000 and IWG 2006 criteria will be held at 12 and 24 weeks of treatment

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Must be 18 years of age or older at the time of screening
* Myelodysplastic Syndrome of the following subtypes : RA, RAS, RCMD, RCMD-RS, RAEB 1, with IPSS score low or intermediate 1 (IPSS score < 1 ) and with anemia defined by Hb < 10 g/dl (with RBC transfusion requirement or not)
* For women of childbearing potential, need for effective contraception throughout the study period.

Exclusion Criteria:

* Intensive Chemotherapy within 3 months before inclusion
* Myelodysplastic Syndrome with IPSS score >1
* Treatment with rHu-Epo or rHu-GCSF within 2 months before inclusion
* EGOG > 3 ;
* Other causes of anemia (eg. , Iron deficiency, vitamin B12 or folic acid, hypothyroidism before correction)
* Uncontrolled arterial hypertension
* Life expectancy less than 6 months
* CMML
* Pregnant or breast feeding female subjects
* Patients with creatinine clearance less than 30ml/min.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2010-06; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Assess the level of haematological response according to IWG 2006 criteria with a pattern of administration of high doses epoetin beta (NeoRecormon ®) for 12 and 24 weeks of treatment | 12 and 24 weeks

CONTACTS AND LOCATIONS:
Locations (31):
- France (31):
  - CHU d'AMIENS, Amiens
  - CH Angers, Angers
  - CH d'Avignon-305 rue Follereau-, Avignon
  - Hopital de la Cote Basque, Bayonne
  - Hôpital Avicenne, Bobigny
  - Hôpital Boulogne Sur Mer, Boulogne-sur-Mer
  - CHU de Brest, Brest
  - CHU Clémenceau, Caen
  - CH René Dubos, Cergy-Pontoise
  - Centre Hospitalier du Mans, Le Mans
  - CHRU Huriez, Lille
  - Hopital Saint-Vincent de Paul-, Lille
  - CHRU de Limoges, Limoges
  - centre hospitalier de Mantes-la-jolie, Mantes-la-Jolie
  - Institut Paoli Calmette, Marseille
  - CHU Brabois, Nancy
  - Hematology Dpt, Hopital de l'Hotel Dieu, Nantes
  - Hôpital Américain de Paris, Neuilly-sur-Seine
  - CHU Archet, Nice
  - Hôpital La Source, Orléans
  - Hôpital Saint Louis, Paris
  - Hôpital Saint-Antoine., Paris
  - Hopital Cochin, Paris
  - Hôpital Jean Bernard, Poitiers
  - Centre Hospitalier de la région d'Annecy, Pringy
  - CHU de Reims, Reims
  - Centre Henri Becquerel, Rouen
  - Centre Hospitalier Universitaire de STRASBOURG, Strasbourg
  - Chu Purpan, Toulouse
  - Hopital Bretonneau, Tours
  - CHU de Bicêtre, Le Kremlin-Bicêtre, Île-de-France Region